CLINICAL TRIAL: NCT06255379
Title: An Open, Single-arm, Multicenter, Prospective Phase II Study of Fuquinitinib Combined With Tegafur Gimeracil Oteracil in the Third-line Treatment of Patients With Advanced Metastatic CRC
Brief Title: Study of Fruquintinib Combined With Tegafur Gimeracil Oteracil in Patients With Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZF-2023-387-01; HMPL-013-SC-CRC102 (Other: Hutchmed)
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Metastasis Colorectal Cancer; Colon Cancer; Rectal Cancer
Keywords: Colorectal cancer; Fruquintinib; Tegafur Gimeracil Oteracil; mCRC
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fuquinitinib +Tegafur Gimeracil Oteracil (Experimental)
  Interventions: Drug: Fuquinitinib+Tegafur Gimeracil Oteracil

INTERVENTIONS:
Drug: Fuquinitinib+Tegafur Gimeracil Oteracil — Fuquinitinib:5 mg once daily, 2 weeks on/1 week off,q3w; Tegafur Gimeracil Oteracil:BSA(body surface area)< 1.2m2,40mg/m2,p.o,bid,2 weeks on/1 week off,q3w; 1.2m2 < BSA （body surface area）< 1.5m2,50mg/m2,p.o,bid,2 weeks on/1 week off,q3w;BSA（body surface area） >1.5m2,60mg/m2,p.o,bid,2 weeks on/1 week off,q3w;

SUMMARY:
This is an Open, Single-arm, Multicenter, Prospective Phase II Study of Fuquinitinib Combined With Tegafur Gimeracil Oteracil in the Third-line Treatment of Patients With Advanced Metastatic CRC

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 75 years of age;
2. Have fully understood and voluntarily sign the ICF for this study (the icf must be signed before any trial-specific procedures are performed);Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure;
3. Histologically and/or cytologically documented metastatic colorectal adenocarcinoma;
4. Refractory to at least second line standard treatment containing fluorouracil, oxaliplatin and irinotecan;
5. At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan or 20mm by conventional CT scan);
6. ECOG performance status of 0-1;
7. Life expectancy ≥ 12 weeks;
8. No previous treatment with vascular endothelial growth factor receptor (VEGFR) inhibitor (TKI);
9. Adequate hepatic, renal, heart, and hematologic functions;
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Any factors that influence the usage of oral administration or any disease or condition that affects drug absorption;
3. Previous treatment with Tegafur Gimeracil Oteracil ;
4. Participated in clinical trials of other drugs within four weeks before enrollment;
5. Received other systemic anti-tumor therapy within 4 weeks before enrollment, including chemotherapy, signal transduction inhibitors, hormone therapy and immunotherapy;
6. International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN;
7. Clinically significant electrolyte abnormalities;
8. Subjected with hypertension that cannot be controlled by drugs, which is specified as: systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg;
9. Unrelieved toxic reactions higher than CTCAE V5.0 grade 1 caused by any previous anti-cancer treatment;
10. Incomplete healing of skin wound, surgical site, traumatic site, severe mucosal ulcer or fracture;
11. Conditions that may cause gastrointestinal bleeding and perforation determined by the researcher;
12. History of arterial thrombosis or deep venous thrombosis within 6 months before enrollment;
13. Stroke and / or transient cerebral ischemia occurred within 12 months before enrollment;
14. Cardiovascular diseases with significant clinical significance;
15. LVEF<50%;
16. Congestive heart failure New York Heart Association (NYHA) grade > 2;
17. Evidence of CNS metastasis;
18. Previous treatment with VEGFR inhibition;
19. Ventricular arrhythmias requiring drug treatment;
20. Proteinuria ≥ 2+ (1.0g/24hr);
21. Coagulation dysfunction, hemorrhagic tendency or receiving anticoagulant therapy;
22. Other malignant tumors in the past 5 years, except skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ;
23. Active infection that is not controlled clinically, such as acute pneumonia, active hepatitis B or hepatitis C;
24. By judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2027-03-21 (Estimated); Study Completion 2027-03-21 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | from randomization up to progressive disease or EOT due to any cause, up to 2 years
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

SECONDARY OUTCOMES:
Objective response rate(ORR) | from randomization up to progressive disease or EOT due to any cause, up to 2 years
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.
Disease control rate(DCR) | from randomization up to progressive disease or EOT due to any cause, up to 2 years
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
Overall survival (OS) | from randomization up to progressive disease or EOT due to any cause, up to 3 years
  OS is the time from enrollment to death due to any cause.
adverse events (AE) | from day 1 of first dosing to 30days after permanent discontinuation of fruquintinib
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No